CLINICAL TRIAL: NCT03034876
Title: Acute Kidney Injury Based on Neutrophil Gelatinase-Associated Lipocalcin (NGAL) in a Pediatric Intensive Care Unit of Tertiary Care Hospital Karachi, Pakistan
Brief Title: Utility of NGAL to Diagnose AKI in Critically Ill Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Anwar ul Haq, Associate Professor, Aga Khan University
Other Study IDs: 4399-Ped-16
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Acute Kidney Injury in Critically Ill Children
Keywords: "Acute Kidney Injury", diagnosis, children, shock
MeSH Terms: conditions — Acute Kidney Injury; Disease; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma of participants will be analyzed for creatinine and Neutrophil Gelatinase-Associated Lipocalcin (NGAL
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute Kidney Injury is common in critically ill children and is associated with high morbidity and mortality in pediatric intensive care unit. The serum creatinine is still a gold standard test for diagnosis of AKI, but it rises after 1 to 3 days of injury . However, Neutrophil Gelatinase-Associated Lipocalcin (NGAL) is an emerging biomarker in identifying AKI at an early stages, which may in future help us in promptly instituting reno-protective interventions like avoidance of nephrotoxic exposure and contrast agents, maintenance of euvolemia and perfusion pressure which will not only preventing kidney from further failing, decrease the use of very expensive and complicated renal supportive therapy like continuous renal replacement therapy (CRRT) as well as in decreasing morbidity and mortality related to AKI.

DETAILED DESCRIPTION:
Introduction:

Acute kidney injury (AKI) is complex disorder affecting the millions of children around the world where approximately 46% of critically ill individual developed acute kidney injury every year (1, 2). An annual incidence of 3.3 cases/100,000 children along with hospital mortality rate of up to 25-50% have reported from developed countries (3) This is even high for developing countries, where annual incidence is 30-50% (4, 5). Furthermore, acute kidney injury leads to significant healthcare use, with cost estimated between 8 billion dollars (4). An early diagnosis is the key to prevent morbidity and mortality related to AKI.

The diagnosis of AKI depends upon elevated serum creatinine level or decrease in urine output . Early detection of AKI is essential. The currently use creatinine clearance (CrCl) is calculated through Schwartz formula. The level of serum creatinine is poor marker for early diagnosis. Because it varies with age, gender, hydration and muscle mass and metabolism. Creatinine never rise until >50% of renal function lost, amount of tubular secretion overestimate at lower GFR, and in acute changes in GFR. During acute changes of GFR in AKI, serum creatinine doesn't accurately depict kidney function until steady state equilibrium has been achieved, which may require several days. There are some biomarker, with high sensitivity and specificity, which can be used as a tool for early detection of AKI, and prevent the burden of mortality and morbidity in intensive care unit (6, 7). Neutrophil gelatinase-associated Lipocalcin (NGAL) recently identified as one of robust marker in AKI (8). Several published reports that plasma NGA is raised in acute kidney injury before rise in serum creatinine (9). A Study conducted by Mishra et al, in US showed that the 2 hours sensitivity is 70% and specificity 94% for NGAL to predict AKI (10). A developed country data showed 84% and 79% sensitivity , and 96% and 90% specificity of NGAL to predict the AKI (2, 11) , (see Annexure 1) . However, there is scarce of information available as plasma NGAL is an early diagnostic marker from Pakistan.

Rationale:

We know that serum creatinine is a gold standard for diagnosis of AKI it is cheaper test to diagnose , but it rises after 1 to 3 days of injury . However, NGAL is a relatively costly test but an emerging biomarker in identifying AKI at an early stages, which may in future help us in promptly instituting reno-protective interventions like avoidance of nephrotoxic exposure and contrast agents, maintenance of euvolemia and perfusion pressure which will not only preventing kidney from further failing, decrease the use of very expensive and complicated renal supportive therapy like continuous renal replacement therapy (CRRT) as well as in decreasing morbidity and mortality related to AKI.

Objective:

To determine the diagnostic accuracy of serum neutrophil gelatinase-associated Lipocalcin (NGAL) , in detection of acute kidney injury by comparing creatinine clearance which is gold standard , in pediatric intensive care unit of Aga khan university hospital Karachi .

Methods:

We will be conducting a prospective observational study in a closed multidisciplinary-cardiothoracic Pediatric Intensive Care Unit (PICU) of Aga Khan University Hospital after approval of Ethical Review Committee.

Operational Definition:

Acute Kidney Injury (AKI): AKI is diagnosed according to pediatric RIFLE criteria. Pediatric RIFLE criteria stratifies AKI when eCrCl decreased by 25 % in first 48hours of PICU.

Shock: Shock is defined by use of vasoactive-inotropic support for at least more than 12 hours to maintain hemodynamics of acutely ill children in PICU for this study.

Neutrophil gelatinase-associated Lipocalcin (NGAL): NGAL is biomarker is measured quantitatively by a rapid , non - competitive Fluorescence Immunoassay (12) . Level of more than 150 mg/dl will be considered as a positive for diagnosis of AKI.

Sample Size Calculation:

If prevalence of AKI in children with shock is 46%, the sensitivity and specificity of plasma NGAL is 0.9 and 0.79 respectively and margin of error is 0.1%, the sample size will be 140 participants.

Participants:

* Inclusion Criteria: All children with either gender aged of 1 month - 16 years who required vasoactive-inotropic drugs on admission and stayed for more than 48 hours in PICU of tertiary care unit of Aga Khan University Hospital, Karachi.
* Exclusion Criteria: All those children who with chronic kidney disease or previous history of renal injury will be excluded

Study Protocol:

The participants who fulfill inclusion and exclusion criteria of the study will be enrolled by daily surveillance of PICU. The informed consent will be obtained from parents or legal guardian. The amount of blood about 1/3rd tea spoon ( 1.5ml ) will be collected from already existing central line without any extra prick of participants at three different time interval of 0 , 12 and 48 hours for plasma-NGAL and serum creatinine test in PICU. Then samples will be sent to main laboratory of our hospital . Blood tests ( NGAL and Serum Creatinine ) expenses will be paid from approved grant of University Research Council . Serum NGAL is measured quantitatively by a rapid , non - competitive Fluorescence Immunoassay (12) . The Triage® NGAL test is a point - of - care , fluorescence - based immunoassay used in conjunction with the Triage Meter (Biosite Inc . ) for the rapid quantitative measurement of NGAL concentration. The serum creatinine will be measured by Jafe's method on ADVIA 1800 Chemistry System (Siemens Healthliners, Germany) , and then creatinine clearance will be calculated by modified Schwartz formula . (19)

Data Collection:

Data variables will be collected on a structured case report form which included demographic variables (age, gender, weight, height), clinical and laboratory variables like admission diagnosis, comorbidities, severity illness score (PRISM III score), use of vasoactive drugs, mechanical ventilation, urine output, fluid balance, serum creatinine and plasma NGAL. The discharge status as alive vs. expired, length of mechanical ventilation and hospitalization and use of renal supportive therapy like peritoneal dialysis will also recorded on case report form.

Outcome:

The primary outcome of this study is to evaluate the level of plasma NGAL in children who is in shock with and without AKI according to RIFLE criteria.

Statistical Analysis:

Data will be entered and analyzed into SPSS V20 (SPSS Inc. Chicago, IL).Normally distributed continuous variables will be reported as mean with standard deviation (SD) and will be compared with student's test. Non-normally continuous distributed data will be reported as medians with interquartile range (IQR) and will be compared with Man Whitney test and Kruskal Wallis test. The categorical data will be reported as proportion and will be compared as Fischer's exact test or Chi-square test. The association between variables will be assessed by Spearman rank order correlation analysis. The diagnostic accuracy of plasma NGAL to predict AKI in children with shock will be defined by calculation of Area Under Curve (AUC) of Receiving Operating Characteristics (ROC) Curves. An AUC of 0.5 is no better than by chance, whereas a value of 1.0 indicates a perfect biomarker. A p-value of <0.05 was considered as statistically significant.

Ethical Consideration:

All data variables will be stored in a password protected computer and strict confidentiality will be maintained.

ELIGIBILITY:
Inclusion Criteria:

All critically ill children who is recieving inotrope in pediatric intensive care unit -

Exclusion Criteria:

* Pre-existing kidney disease
* Chronic kidney disease

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All critically ill children admitted in pediatric intensive care unit and receiving inotrope
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute Kidney Injury | within 24 hour
  serum will sent to plasma any time of day and test will run once a day

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rustagi RS, Arora K, Das RR, Pooni PA, Singh D. Incidence, risk factors and outcome of acute kidney injury in critically ill children - a developing country perspective. Paediatr Int Child Health. 2017 Feb;37(1):35-41. doi: 10.1080/20469047.2015.1120409. Epub 2016 Jan 9. PMID 26752169
- [Background] Naik S, Sharma J, Yengkom R, Kalrao V, Mulay A. Acute kidney injury in critically ill children: Risk factors and outcomes. Indian J Crit Care Med. 2014 Mar;18(3):129-33. doi: 10.4103/0972-5229.128701. PMID 24701061
- [Background] Waikar SS, Bonventre JV. Biomarkers for the diagnosis of acute kidney injury. Nephron Clin Pract. 2008;109(4):c192-7. doi: 10.1159/000142928. Epub 2008 Sep 18. PMID 18802367
- [Background] Haase M, Bellomo R, Devarajan P, Schlattmann P, Haase-Fielitz A; NGAL Meta-analysis Investigator Group. Accuracy of neutrophil gelatinase-associated lipocalin (NGAL) in diagnosis and prognosis in acute kidney injury: a systematic review and meta-analysis. Am J Kidney Dis. 2009 Dec;54(6):1012-24. doi: 10.1053/j.ajkd.2009.07.020. Epub 2009 Oct 21. PMID 19850388
- [Background] Doi K, Negishi K, Ishizu T, Katagiri D, Fujita T, Matsubara T, Yahagi N, Sugaya T, Noiri E. Evaluation of new acute kidney injury biomarkers in a mixed intensive care unit. Crit Care Med. 2011 Nov;39(11):2464-9. doi: 10.1097/CCM.0b013e318225761a. PMID 21705884